CLINICAL TRIAL: NCT05086302
Title: A Postmarket Study for Continuing Evaluation and Periodic Reporting of the Safety and Effectiveness of the Spatz3 Intragastric Balloon
Brief Title: Spatz3 Adjustable Balloon System® (Spatz3) Post Approval Study
Status: Completed | Type: Observational
Sponsor: Spatz FGIA, Inc (Other)
Responsible Party: Sponsor
Other Study IDs: Spatz3-PAS
Record Dates: First submitted 2021-10-19; First posted 2021-10-20 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 56 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
A prospective, Multicenter open-label post approval trial for adults with a Body Mass Index (BMI) of 35.0-40.0 kg/m2 or a BMI of 30.0 to 34.9 kg/m2 with one or more major obesity-related comorbid conditions who have failed to achieve and maintain weight-loss with a supervised weight control program.

The study aims to demonstrate that the safety of the device in the post market setting is comparable to what was observed in the US pivotal study.

DETAILED DESCRIPTION:
The purpose of the study is to demonstrate that the safety of the device in the postmarket setting is comparable to what was observed in the US pivotal study and to more accurately determine the rates of certain serious adverse events so that this information can be used to inform patient labeling.

Subjects in the open label, multi-center study will receive dietary/exercise counseling plus the Spatz3 Adjustable Balloon System for 32 weeks.

Eligible subjects will undergo endoscopy and those without endoscopic contraindications will be implanted with the Spatz3 Adjustable Balloon System for 32 weeks. All subjects will follow a 1000-1200 kcal/day-deficit diet during their participation in the study.

At 18 weeks ±4 weeks, subjects will be evaluated, and those that meet the criteria will undergo an adjustment procedure wherein the balloon volume will be increased to achieve extra weight loss. The balloon adjustment procedure is done with an endoscopy procedure under the same sedation as the implantation procedure.

At the end of the 32-week treatment period, all subjects who lost at least 5% Total Body Weight Loss (TBWL) prior to device removal will be followed for an additional 6 months. In addition, patients with device- and/or procedure-related adverse events will be followed until resolution of the event

ELIGIBILITY:
Inclusion Criteria:

1. Age 22 - 65
2. BMI ≥ 35 and <40 kg/m2 or BMI of 30 to 34.9 kg/m2 with one or more major obesity- related comorbid conditions
3. Willingness to comply with the substantial lifelong dietary restrictions required by the procedure
4. History of obesity (BMI ≥ 30) for at least 2 years
5. History of failure with non-surgical weight loss methods
6. Willingness to follow protocol requirements, including signed informed consent, routine follow-up schedule, completing laboratory tests, completing diet counseling
7. Residing within a reasonable distance from the investigator's office and able to travel to the investigator to complete all routine follow- up visits
8. Ability to give informed consent
9. Women of childbearing potential (i.e., not post-menopausal or surgically sterilized) must agree to use adequate birth control methods. Acceptable birth control methods are limited to hormonal contraceptives (oral, flexible vaginal ring, skin patch, injection), diaphragms, IUDs, condoms with or without spermicide, and voluntary abstinence. Should a treatment arm subject become pregnant during the implantation period, the balloon will be extracted during the second trimester - the timing of which will be determined via consultation with the subject's obstetrician.

Exclusion Criteria:

1. Prior surgery involving the esophagus, stomach, and duodenum or bariatric surgery.
2. Prior open or laparoscopic bariatric surgery.
3. Prior surgery of any kind on the esophagus, stomach, duodenum or any type of hiatal hernia surgery.
4. Any inflammatory disease of the gastrointestinal tract including esophagitis, Barrett's esophagus, gastric ulceration, duodenal ulceration, cancer or specific inflammation such as Crohn's disease
5. Potential upper gastrointestinal bleeding conditions such as esophageal or gastric varices, congenital or acquired intestinal telangiectasis, or other congenital anomalies of the gastrointestinal tract such as atresias or stenoses.
6. A gastric mass.
7. A hiatal hernia > 2cm or severe or intractable gastro-esophageal reflux symptoms.
8. Acid reflux symptoms to any degree that require more than one medication for symptom control.
9. A structural abnormality in the esophagus or pharynx such as a stricture or diverticulum that could impede passage of the balloon alongside the endoscope.
10. Achalasia or any other severe esophageal motility disorder that may pose a safety risk during the removal of the device
11. Severe coagulopathy.
12. Insulin-dependent diabetes (either Type 1 or Type 2) or a significant likelihood of requiring insulin treatment in the following 12 months.
13. Subjects with any serious health condition unrelated to their weight that would increase the risk of endoscopy
14. Chronic abdominal pain
15. Motility disorders of the GI tract such as gross esophageal motility disorders, gastroparesis or intractable constipation
16. Hepatic insufficiency or cirrhosis
17. Serious or uncontrolled psychiatric illness or disorder that could compromise patient understanding of or compliance with follow up visits and removal of the device after 8 months.
18. Alcoholism or drug addiction.
19. Patients unwilling to participate in an established medically-supervised diet and behavior modification program, with routine medical follow-up.
20. Patients receiving daily prescribed treatment with aspirin, anti-inflammatory agents, anticoagulants or other gastric irritants.
21. Patients who are unable or unwilling to take prescribed proton pump inhibitor medication for the duration of the device implant.
22. Patients who are known to have, or suspected to have, an allergic reaction to materials contained in the system.
23. Patients who have BOTH:

    1. A previous history of a serotonin syndrome AND
    2. currently taking any drug known to affect the levels of serotonin in the body [e.g., selective serotonin reuptake inhibitors (SSRIs), serotonin-norepinephrine reuptake inhibitors (SNRIs), monoamine oxidase inhibitors (MAOIs)].
24. Patients who are pregnant or breast-feeding.
25. Subjects with Severe cardiopulmonary disease or other serious organic disease which might include known history of coronary artery disease, Myocardial infarction within the past 6 months, poorly controlled hypertension, required use of NSAIDs
26. Subjects who have tested positive for H. Pylori, and who have not yet been treated.
27. Subjects taking medications on specified hourly intervals that may be affected by changes to gastric emptying, such as anti-seizure or anti-arrhythmic medications
28. Subjects who are taking corticosteroids, immunosuppressants, and narcotics
29. Subjects who are taking diet pills
30. Use of an intragastric device prior to this study due to the potential increase in risk associated with implantation of a balloon in a previously instrumented and possibly scarred stomach.
31. Participation in any clinical study which could affect weight loss within the past 6 months due to the potential to confound findings.
32. Symptomatic congestive heart failure, cardiac arrhythmia or unstable coronary artery disease.
33. Pre-existing respiratory disease such as chronic obstructive pulmonary disease (COPD), pneumonia or cancer.
34. Diagnosis of autoimmune connective tissue disorder (e.g. lupus, erythematous, scleroderma) or immunocompromised.
35. Life expectancy less than 1 year or severe renal, hepatic, pulmonary or other medical condition, in the opinion of the investigator because of an increased risk profile.
36. Specific diagnosed genetic or hormonal cause for obesity such as untreated hypothyroidism or Prader Willi syndrome
37. Eating disorders including night eating syndrome (NES), bulimia, binge eating disorder, or compulsive overeating
38. Known history of endocrine disorders affecting weight

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with a Body Mass Index (BMI) of 35.0-40.0 kg/m2 or a BMI of 30.0 to 34.9 kg/m2 with one or more major obesity-related comorbid conditions who have failed to achieve and maintain weight-loss with a supervised weight control program.
Sampling Method: Non-Probability Sample
Enrollment: 537 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Events (SAEs) | 32 weeks
  The primary study endpoint is to demonstrate that the rate of device or procedure related SAEs is less than 8% at 8 months

SECONDARY OUTCOMES:
Percentage of Total Body Weight Loss (%TBWL) | 32 weeks
  The secondary study endpoint is to demonstrate that the mean percent TBL in the effectiveness cohort is not less than 11% at 32 weeks.
Mean %TBL and percent excess weight loss (EWL%) | 56 weeks
  Mean %TBL and percent excess weight loss (EWL %) at 56 weeks in subjects who lost at least 5% TBL at 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Brooks, MD, Study Director — Spatz FGIA, Inc
Locations (22):
- United States (20):
  - Carson D Liu MD Medical Corp, Marina del Rey, California
  - JSAPA, Jupiter, Florida
  - Formation, Tampa, Florida
  - True You Weight Loss (Atlanta), Atlanta, Georgia
  - Gastro Center of Maryland, Columbia, Maryland
  - The Silhouette Clinic, Germantown, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Reveal Weight Loss, Livingston, New Jersey
  - Weight Loss and Wellness Center, Livingston, New Jersey
  - New Jersey Bariatric Center, Springfield, New Jersey
  - New York Bariatric Group - Wayne Location, Wayne, New Jersey
  - Steven Batash, M.D., P.C., New York, New York
  - True You Weight Loss, Cary, North Carolina
  - Atlantic Medical Group, Kinston, North Carolina
  - JourneyLite Physicians, Cincinnati, Ohio
  - NRHS Journey Clinic, Norman, Oklahoma
  - Basin Surgical, Midland, Texas
  - Endoscopic Wellness Center of America, Reston, Virginia
  - Advanced Gastroenterology & Hepatology of Greater Washington, Vienna, Virginia
  - Transform Weight Loss, Seattle, Washington
- Puerto Rico (2):
  - FRC Gastro, Bayamón, Puerto Rico
  - GI Offices of Dr. Rodriguez and Dr. Osorio, Bayamón, Puerto Rico